CLINICAL TRIAL: NCT02887742
Title: Epidemiologic Study and Impact Study of a Dialysis Solution Change on the Electrocardiographic Profile of Patient
Acronym: QT_DIAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: QT-DIAL (10.014)
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2016-08

CONDITIONS: Haemodialysis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiologic Study and Impact Study of a Dialysis Solution Change on the Electrocardiographic Profile of Patient

ELIGIBILITY:
Inclusion Criteria:

* >18
* patient under haemodialysis treatment
* patient not objecting to study

Exclusion Criteria:

* Patient with known cardiac arrythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialysed patients from two nephrology centers.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Description of all the cardiologic abnormalities | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le meur, MD PhD, Study Director — University Hospital, Brest
Locations (2):
- France (2):
  - AUB, Brest
  - CHU Brest, Brest